CLINICAL TRIAL: NCT03894410
Title: Real World Study of Lapatinib Among Metastatic Breast Cancer Patients in Clinical Practice: a Multicenter, Retrospective Study
Brief Title: Real World Study of Lapatinib Among Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-6
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: HER2; Lapatinib
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Continuing Lapatinib: Patients continued using treatment containing Lapatinib after progression on Lapatinib.
- Change HER-2 treatment: Patients changed to another HER-2 targeted treatment after progression on Lapatinib (ado-trastuzumab emtansine, trastuzumab, etc.).
- Lapatinib plus capetabine: Patients used lapatinib plus capetabine.
- Lapatinib plus Trastuzumab and one chemotherapy: Patients used lapatinib plus trastuzumab and one chemo regimen.

SUMMARY:
A multicenter, retrospective, real world study of Lapatinib among Metastatic Breast Cancer (MBC) Patients in Clinical Practice.

DETAILED DESCRIPTION:
This study collected patients used Lapatinib-base therapy among MBC, and tried to figure out if there was difference between single anti-Her2 treatment and dual anti-Her2 treatment. Furthermore, this study investigated the treatment after Lapatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated with Lapatinib between June 2014 to June 2018.
* Patients experienced progression on prior trastuzumab-containing regimens and a taxane.
* Complete medical history was available.

Exclusion Criteria:

* Medical history was incomplete.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided